CLINICAL TRIAL: NCT00169871
Title: Hs-CRP as Clinical Marker of Inflammatory Atherogenic Dyslipidemia
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: AstraZeneca (Industry)
Other Study IDs: DC-452-0011
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2006-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The objective of this proposal is to study the applicability of the hs-CRP assay in the assessment of CV risk in daily clinical conditions where hyperlipidemic population with or without CHD are currently evaluated.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the major cause of death in the developed world. Cholesterol screening has been used as a tool to identify individuals who are at increased risk of developing future coronary events, but almost one-half of patients who develop myocardial infarction have either normal or only moderately increased serum cholesterol concentrations. In the last years, experimental and clinical evidence has demonstrated that atherosclerosis is not simply a disease of lipid deposits. Rather, there is growing recognition that CHD has an inflammatory component which plays a critical role in the arterial plaque rupture that triggers most episodes of coronary thrombosis. In the last years, C-reactive protein (CRP), an exquisitely sensitive marker of systemic inflammation, has emerged as a powerful predictor of cardiovascular diseases, in particular of CHD, beyond what can be estimated by traditional risk factors. The availability of high-sensitivity (hs) CRP assays has enabled the detection of even low-grade inflammatory responses that have previously been regarded as clinically not meaningful. However, for hs-CRP to make the transition from epidemiological and clinical research to the routine clinical setting, several important issues must be satisfactorily addressed.

Therefore, the overall objective of this proposal is to study the applicability of the hs-CRP assay in the assessment of CV risk in daily clinical conditions where hyperlipidemic population with or without CHD are currently evaluated and to evaluate hs-CRP response to statins.

ELIGIBILITY:
Inclusion Criteria:

* metabolically stable in the last 3 months for weight (+/- 1 kg), lipid profile (+/- 15 % variability), infection (no symptoms for viral or bacterial illness), inflammation (absence of nonspecific symptoms for arthritis, normal blood sedimentation and protein electrophoresis for acute phase reactants) and no change of usual habits (ex. diet/exercise) or medications (ex. drugs)
* CHD patients will have to be stable (based on cardiac symptoms and ECG) during the last 3 months and diabetic patients will be required to have stable glycemia (HbA1c < 7,5 %) in the last 6 months.

Exclusion Criteria:

* history of drug or alcohol abuse
* uncontrolled liver, thyroid or kidney functions
* other drugs known to affect lipid levels or insulin resistance (antiprotease inhibitors, oral contraceptives...)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-03; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bergeron, MD MSc FRCPC, Principal Investigator — CHUL Research Center
Locations (1):
- Lipid Research Center, CHUL Research Center, Sainte-Foy, Quebec, Canada